CLINICAL TRIAL: NCT06503198
Title: Virtual, Innovative, Postsurgical Care To Optimize Return Home for Older People With frailtY: the VICTORY Randomized Trial
Brief Title: The VICTORY Trial: Virtual, Innovative, Postsurgical Care To Optimize Return Home for Older People With frailtY
Acronym: VICTORY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230610-01T
Record Dates: First submitted 2024-06-24; First posted 2024-07-16 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Surgery; Frailty
MeSH Terms: conditions — Frailty | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Individual patient, parallel-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The VICTORY Trial is a multicenter, innovative clinical trial using an individual patient, parallel-arm randomized controlled trial design of 1,000 older patients living with frailty being discharged from hospital after elective surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Care (Experimental): Intervention group participants will be enrolled in a PVC program prior to admission, including receipt of a cellular-enabled tablet and Cloud DX remote monitoring equipment.
  Through Cloud DX remote monitoring technology, intervention group participants will receive the following intervention: remote automated monitoring, frailty-tailored daily symptom survey, Katz Index of Independence in Activities of Daily Living survey, FAM-CAM survey, Virtual RN assessment, medications.
  Interventions: Behavioral: Virtual care
- Standard Care (No Intervention): The standard care group will receive their post-hospital discharge management in alignment with standard of care at the hospital where they had surgery.

INTERVENTIONS:
Behavioral: Virtual care — Through Cloud DX, intervention group participants will receive:
  Remote Automated Monitoring: measurement of: blood pressure, heart rate, respiratory rate, oxygen saturation, temperature and weight.
  Frailty-tailored daily symptom survey: The recovery survey consists of questions related to infection, bleeding, pain, appetite, dehydration, appetite, syncope and falls.
  The tablet will prompt the participant to complete a Katz Index of Independence in Activities of Daily Living (IADL) survey. The FAM-CAM survey will also be pushed by Cloud DX to be completed.
  Virtual RN assessment: a virtual RN assessment will be scheduled at a minimum of every 2 days for the first 7 days. The virtual RN will also perform the 4AT Delirium Assessment.
  Medications: the virtual RN will undertake medication review and reconciliation. In addition, they will provide counselling regarding analgesic support and monitor for drug interactions.
  Arms: Virtual Care

SUMMARY:
Canadian hospitals continue to struggle with severe emergency department and hospital bed capacity shortages. Maximizing bed availability and minimizing emergency department and urgent-centre visits by providing patients with alternative options to care is an important part of the solution. Surgical patients with frailty are at high risk of requiring subsequent acute-hospital care. The VICTORY trial will answer an important question that will inform how to improve care for surgical patients with frailty by determining the effect of virtual care with CloudDX technology compared to standard care to see if it can result in an increase in the number of days alive and at home that older people with frailty experience after planned surgery.

DETAILED DESCRIPTION:
Background: Each year, >130,000 older Canadians living with frailty have major, inpatient surgery. The presence of frailty, a multidimensional state of vulnerability, is strongly associated with adverse outcomes. Compared to similar patients without frailty, surgical patients with frailty experience a 2- to 5-fold adjusted increase in the odds of mortality, complications, patient-reported disability, length of stay, readmissions and non-home discharge. However, despite the growing number of patients with frailty presenting for surgery each year, a recent systematic review from our team demonstrates that there are no evidence-based, frailty-specific interventions available to drive improvements in outcomes for this vulnerable population. A promising intervention to support independence and maintain older people at home after surgery is Virtual Recovery After Surgery (VRAS), an innovative multidisciplinary program that has been providing post-discharge remote monitoring and virtual care for surgical patients since 2021. Patients receive virtual care from the VRAS nursing and anesthesiologist team following surgical discharge, facilitated by Cloud DX software and monitoring equipment. Based on our team's joint expertise in frailty and Postoperative Virtual Care (PVC), the investigators have identified: 1) a crucial gap in care expressed by older patients with frailty (the need for support and continuity of care via telehealth resources to support transition of care to their homes), and 2) an intervention that could directly fill this gap (frailty tailored PVC).

Overarching Aim: The objective of the VICTORY Trial is to determine the effect of virtual care with CloudDX technology compared to standard care to see if it can result in an increase in the number of days alive and at home that older people with frailty experience in the 30 days after planned surgery. A secondary aim is to estimate the probability that enrollment in a frailty-tailored PVC program will reduce healthcare resource use and improve patient-reported outcomes and safety.

Methods:

Design, setting and participants: The VICTORY Trial is a multicenter, innovative clinical trial using an individual patient, parallel-arm randomized controlled trial design of 1,000 older patients living with frailty being discharged from hospital after elective surgery.

People ≥60 years old with frailty having elective surgery will be included.

Intervention: Patients randomized to the PVC program will be monitored at home by virtual nurses for at least 7 days after hospital discharge. Participants will be provided with a hospital-to-home kit that contains the following technologies: tablet computer (with stand), wrist-based blood pressure cuff (for blood pressure, pulse and breathing rate), finger worn pulse oximeter (for measuring oxygen levels), thermometer (for temperature) and weigh scale (to monitor weight). Monitoring will include video visits with a nurse on post-discharge days 1, 3, 5 and 7 and every other day until post-discharge day 14 if needed. Patients will be asked to complete a daily survey that will include questions about any symptoms they may be experiencing, their independence/dependence with activities of daily living, and their experience with the PVC program. Depending on the patient's recovery (including the assessments and surveys described), patients may receive information electronically on how to manage certain challenges (i.e., confusion, not eating enough), their care may be escalated to a physician, or they may be instructed to come to the hospital.

Outcomes and sample size: The primary outcome is the number of days that each patient spends alive and at home following surgery. Secondary outcomes are: resource use (index length of stay, readmission, total hospital days, emergency department visits, time to first acute hospital care, cost of care), patient-centered outcomes (delirium (4AT), quality of life (EQ- 5D-5L), pain interference (PROMIS), satisfaction (likelihood to recommend), goal attainment, and overall quality of transitional care received), safety (medication issues, incidence of post-discharge falls).

Based on trial simulations, the investigators estimate that the most likely number of participants required will be 1000 (500 per arm), which is adequate to achieve at least 90% power to declare superiority (defined as probability of any benefit = 99% (P(Odds Ratio (OR)>1) = 99%) when the effect size, expressed as an OR from a cumulative logistic model, is 1.5 and the control group number of days alive at home within 30 days is 16.

Expertise: Our team features multidisciplinary clinical and methodological experts, nationally representative knowledge users and patient representatives.

Expected outcomes: The VICTORY Trial will: 1) advance the practice of PVC using evidence-based, frailty-tailored approaches; 2) evaluate this frailty-tailored PVC intervention in direct partnership with patients; and 3) produce robust, potentially practice-changing research using innovative clinical trial methodologies that will inform implementation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 60years
2. Diagnosis of frailty (Clinical Frailty Score >4)
3. Elective surgery
4. Fluent in English

Exclusion Criteria:

1. Preoperative institutional residence
2. Planned postoperative non-home discharge (i.e. rehabilitation or convalescence)
3. Patient unable to interact with virtual care and/or technology
4. Cognitive impairment preventing ability to provide independent informed consent to surgery and the trial
5. Patient lives in an area without cellular or internet service

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of days each patient spends alive and at home following surgery | 30 days
  This validated, patient-centered outcome is calculated as the sum of all days alive within 30-days of surgery minus any days spent in hospital (index or readmission), rehabilitation, or nursing home/long term care centers. Death will be assigned a '-1' value; those surviving 30-days will be assigned an outcome value of their count of days alive and at home

OTHER OUTCOMES:
Resource use- Index length of stay | 30 days
  Count of days from date of surgery to hospital discharge will be documented
Resource use- Readmission | 30 days, 1 year
  Any acute care hospitalization after index hospital discharge and within 30-days and 365-days of surgery will be documented
Resource use- Readmission length of stay | 30 days
  Sum of total counts of days from start of new acute care admission to discharge where the New admissions occurring within 30 days of index surgery will be documented
Resource use- 30-day total hospital days | 30 days
  Count of all days spent in an acute care hospital from surgery to 30-days after surgery will be documented
Resource use- Number of Emergency Department visits | 30 days, 1 year
  Count of Emergency Department visits occurring between index surgery and 30-days and 365-days after surgery will be documented
Resource use- Time to first acute hospital care | 30 days
  Count of days from index surgical admission discharge to first Emergency Department visit or readmission will be documented
Resource use- Costs of care | 30 days, 1 year
  For Ontario patients, standardized case costing methods will be used to estimate total health system costs from date of surgery to 30-days and 365-days after surgery
Patient-centered- Delirium (4AT) | Days 1 and 3 post-discharge
  Captured using the UltraBrief, a separate delirium screening tool from the 4AT Confusion Assessment Methods utilized as part of the intervention delirium screening. A score of 4 or more suggests delirium but is not diagnostic. A score of 1-3 suggests cognitive impairment and more detailed cognitive testing and informant history-taking may be indicated. A score of 0 does not definitively exclude delirium or cognitive impairment: more detailed testing may be needed depending on the clinical context.
Overall quality of transitional care received | 30 days
  Using the Ideal Transitions in Care (ITC) Framework, which has 10 domains to consider to ensure safe transitions of care. Number of domains will be reported.
Quality of life (EQ- 5D-5L) | 30 days, 90 days
  This is a well-validated instrument with Canadian valuation statistics and national implementation used to measure health-related quality of life after surgery and to inform incremental cost per quality-adjusted life year gained. Participants are asked to select one answer under each domain (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Responses range from having no problems with a particular domain to being unable to engage in that particular domain. Participants are asked to identify on a scale of 0-100 how good or bad their health is on that given day (0 being worst health they can imagine, 100 being best health they can imagine).
Pain interference (PROMIS) | 30 days, 90 days
  The 6-item Short Form 6b V1.0 will be used to capture interference of pain. Item-levels are scored numerically for an individual's response to each question. Higher scores means more of the concept being measured. The lowest raw score is 6 and the highest raw score is 30.
Satisfaction (Likelihood to Recommend) | 30 days
  Patients will complete the 'Likelihood to recommend' question, reflecting on a 10-point scale their likelihood to recommend their postoperative transitional care experience
Personalized goal attainment | 30 days, 90 days
  A method of evaluating the extent to which patient's individual goals are achieved in the course of an intervention, previously used in rehabilitation studies for older adults with frailty, using an 11-point Likert scale; this outcome directly aligns with the 5th geriatric 'M' (matters most) where participants report the most important benefit from surgery and rate the achievement of the goal on a scale from worse than before surgery to much better than I expected after surgery
Safety- Incidence of post-discharge falls | 30 days
  Falls post-discharge
Safety- Medication issues using the Treatment Satisfaction Questionnaire for Medications (TSQM) scale | Day of discharge from program post-surgery (assessed up to day 6)
  The virtual registered nurse will undertake medication review and reconciliation on day 1 and day of discharge from program. In addition, they will provide counselling regarding analgesic support and monitor for drug interactions. Questions from the TSQM scale will be administered. The degree to which medication side effects affected overall satisfaction will be reported on a scale from extremely satisfied to not at all. How satisfied or dissatisfied the participant is with the medications will be reported on a scale from very satisfied to very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Aucoin, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data, including data dictionaries, will be available. This includes individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices). The Study Protocol, Statistical Analysis Plan and Informed Consent Form will also be made available. Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data. Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.
Supporting Information: SAP
Time Frame: Data will be available beginning 3 months and ending 5 years following article publication of one year follow up data.
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data can be used to achieve aims in a proposed proposal or for individual participant data meta-analysis. Proposals should be directed to the Principal Investigator. To gain access, data requestors will need to sign a data access agreement. Data will be shared via an appropriate 3rd party website that is consistent with ethical and health privacy compliant legislation at the time of study conclusion.